CLINICAL TRIAL: NCT05518630
Title: An Investigation of Nomothetic Versus Idiographic Assessment in Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 20220516
Record Dates: First submitted 2022-08-16; First posted 2022-08-26 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis; Vulvodynia; Fibromyalgia
Keywords: Endometriosis; Vulvodynia; Fibromyalgia; Psychological flexibility
MeSH Terms: conditions — Endometriosis; Vulvodynia; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Nomothetic Versus Idiographic Assessment in Chronic Pain — Participants with either endometriosis, vulvodynia, and/or fibromyalgia will answer a twice-daily diary for 42 days and a short weekly diary six times in total. In addition, they will answer two longer surveys at the start and at the end of the 42 days. These questionnaires ask about psychological flexibility, depression, catastrophizing, and pain interference. The data collected is only observational and does not include any intervention.

SUMMARY:
Endometriosis, vulvodynia, and fibromyalgia are chronic pain conditions that cause great suffering. Despite the significant prevalence of all three conditions, they are receiving relatively little attention in psychological treatment research. Despite the popularity of methods that rely on aggregated group data, such as randomized controlled trials (RCTs), concerns have been raised in recent years about the generalizability of results from these methods to the individual level - group-to-individual generalizability. Since psychological treatments in the clinic are focused on enhancing the well-being of a specific individual this might affect how researchers should study these conditions. The current project aims to investigate: (a) item suitability for daily assessment of psychological variables, (b) group-to-individual generalizability in outcome measures frequently used in psychological studies and treatments of chronic pain, (c) relations over time between process and outcome variables, and (d) possible differences in results obtained across three pain conditions.

DETAILED DESCRIPTION:
Endometriosis, vulvodynia, and fibromyalgia are chronic pain conditions that cause great suffering. The pain conditions are associated with suffering both psychologically and physically. However, knowledge about these conditions is scarce.

The present study aims to investigate the relationship between pain intensity, psychological flexibility, pain functioning, catastrophizing, and depressive symptoms in people with endometriosis, vulvodynia, and fibromyalgia. The investigators want to investigate how these factors relate to each other over time, but also whether there is a difference between people who are in contact with health care for these conditions and those who are not, and whether there is a difference depending on which of the included pain conditions one has.

Another aim of the project is to investigate whether the variables the investigators intend to measure meet the criteria for group-to-individual generalizability, meaning that group means and correlation coefficients based on aggregated group data also apply to individuals and that it is reasonable to draw conclusions about individuals from group data. Many psychological variables do not meet the criteria for this type of generalizability. By examining whether the results from variables can be generalized from a group level to an individual level, the investigators will gain clues about how much individualization is required in future research, assessments, and treatments for the pain conditions included in the current project.

In order to investigate group-to-individual generalizability, the project requires a large sample of participants to obtain group averages but also a large number of repeated measurements over a longer period of time for each participant. Repeated measurements from each individual are planned to be carried out to obtain individual mean values, in order to compare this with the group data. A diary will be created which is intended to be used daily, and a further aim of this study is to evaluate whether this diary is valid to use for future studies in these pain conditions.

On the first day of the study, participants will complete forms collecting demographic and background information, including information about the participants' pain.

On the first as well as the last day, information will also be collected from standardized questionnaires, including the Multidimensional Psychological Flexibility Inventory (MPFI), Patient Health Questionnaire-9 (PHQ-9), Brief Pain Inventory (BPI), and Pain Catastrophizing Scale (PCS).

On the second day of the study, participants will start to fill in twice daily measures at fixed times, and with a 12-hour interval between these two daily measurements. These are based on an ecological momentary assessment approach (EMA), where frequently repeated measurements are taken in the natural environment of the research subjects and where the time that participants have to think back on when answering is kept short. Using EMA, the within-individual variation can be easily monitored over time. The daily measurements will be collected for 42 days. The measurements consist of items from MPFI, BPI, PHQ-2, and PCS. In addition, two items are developed by the research team to assess sexual functioning and energy levels.

Participants will also fill out a weekly diary administered six times in total. The weekly diary consists of three items asking the participant to rate the previous week, and indicate whether something out of the ordinary has happened.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Reporting diagnoses of endometriosis, vulvodynia, or fibromyalgia
* The pain condition present persistently or recurrently during ≥ 3 months
* Access to an internet-enabled smartphone/tablet
* Fluent in written Swedish

Exclusion criteria:

- Planned surgery during the upcoming 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People reporting diagnoses of endometriosis, vulvodynia, or fibromyalgia.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Psychological Flexibility Inventory (MPFI) - Psychological Inflexibility subscale | Measured immediately following participant consent to undertake survey
  A 30-item measure reflecting all facets of psychological inflexibility, namely: experiential avoidance, lack of contact with the present moment, self as content, fusion, lack of contact with values, and inaction. The minimum score is an average of 1 across the 30 items, and the maximum score is 6 across the 30 items. It can also be scored on a facet level with a minimum score of 1 and a maximum score of 6 for the individual facet scored. A higher average score indicates higher psychological inflexibility.
Multidimensional Psychological Flexibility Inventory (MPFI) - Psychological Inflexibility subscale | Six weeks after participant consent
  A 30-item measure reflecting all facets of psychological inflexibility, namely: experiential avoidance, lack of contact with the present moment, self as content, fusion, lack of contact with values, and inaction. The minimum score is an average of 1 across the 30 items, and the maximum score is 6 across the 30 items. It can also be scored on a facet level with a minimum score of 1 and a maximum score of 6 for the individual facet scored. A higher average score indicates higher psychological inflexibility.
Psy-Flex | Measured immediately following participant consent to undertake survey
  A 6-item measure assessing all facets of psychological flexibility using one item per facet. The minimum score is 6 and the maximum score is 30. Higher scores indicate higher psychological flexibility.
Psy-Flex | Six weeks after participant consent
  A 6-item measure assessing all facets of psychological flexibility using one item per facet. The minimum score is 6 and the maximum score is 30. Higher scores indicate higher psychological flexibility.
Patient Health Questionnaire-9 (PHQ-9) | Measured immediately following participant consent to undertake survey
  A nine-item measure on symptoms of depression, with a minimum score of 0 and a maximum score of 27. Higher scores indicate higher levels of depression. The scale also includes an additional item regarding how the depressive symptoms have interfered with everyday functioning. Higher scores indicate higher levels of everyday interference.
Patient Health Questionnaire-9 (PHQ-9) | Six weeks after participant consent
  A nine-item measure on symptoms of depression, with a minimum score of 0 and a maximum score of 27. Higher scores indicate higher levels of depression. The scale also includes an additional item regarding how the depressive symptoms have interfered with everyday functioning. Higher scores indicate higher levels of everyday interference.
Pain Catastrophizing Scale (PCS) | Measured immediately following participant consent to undertake survey
  A 13-item measure assessing the level of catastrophizing when in pain. Includes three main factors; rumination, magnification, and helplessness. The minimum score is 0 and the maximum score is 52. Higher scores indicate higher levels of pain catastrophizing.
Pain Catastrophizing Scale (PCS) | Six weeks after participant consent
  A 13-item measure assessing the level of catastrophizing when in pain. Includes three main factors; rumination, magnification, and helplessness. The minimum score is 0 and the maximum score is 52. Higher scores indicate higher levels of pain catastrophizing.
Brief Pain inventory - short form (BPI-SF) | Measured immediately following participant consent to undertake survey
  For this study, two items on pain severity (one regarding average pain severity during the last week and one regarding pain severity at the current moment) and ten items on pain interference will be used. Three out of the ten pain interference items, exploring how pain interferes with sexual activities, enjoyment of sex, and feelings of being rested, have been created and added by the research team. The two pain severity items are each scored from 0 to 10, with 0 indicating the least amount of pain and 10 indicating the highest amount of pain. The original seven pain interference items are each scored in the same way, but can also together generate an average score, with the minimum average score then being 0 and the maximum average score being 10. A higher score indicates a higher level of pain interference. The three pain interference items created by the research team are scored in the same way.
Brief Pain inventory - short form (BPI-SF) | Six weeks after participant consent
  For this study, two items on pain severity (one regarding average pain severity during the last week and one regarding pain severity at the current moment) and ten items on pain interference will be used. Three out of the ten pain interference items, exploring how pain interferes with sexual activities, enjoyment of sex, and feelings of being rested, have been created and added by the research team. The two pain severity items are each scored from 0 to 10, with 0 indicating the least amount of pain and 10 indicating the highest amount of pain. The original seven pain interference items are each scored in the same way, but can also together generate an average score, with the minimum average score then being 0 and the maximum average score being 10. A higher score indicates a higher level of pain interference. The three pain interference items created by the research team are scored in the same way.
Endometriosis Health Profile - 5 (EHP-5) | Measured immediately following participant consent to undertake survey
  A five-item measure assessing quality of life in people with endometriosis. Each item is scored on a four-point scale. The minimum score is 0, and the maximum score is 100. A higher score indicates worse health status. The measure is only administered to participants responding that they suffer from endometriosis.
Endometriosis Health Profile - 5 (EHP-5) | Six weeks after participant consent
  A five-item measure assessing quality of life in people with endometriosis. Each item is scored on a four-point scale. The minimum score is 0, and the maximum score is 100. A higher score indicates worse health status. The measure is only administered to participants responding that they suffer from endometriosis.
Brief Pain inventory - short form (BPI-SF) | Six weeks
  An eight-item questionnaire. One item measuring current pain intensity and seven items measuring pain interference on general activity, mood, sleep, feeling of being rested, relations with other people, enjoyment of life, and enjoyment of sex. The two items measuring pain interference on feelings of being rested and enjoyment of sex are developed by the research team. Item assessing sleep is administered once per day in the morning, and the item assessing feelings of being rested is administered once per day in the evening. Pain intensity is scored from 0 to 10, with 0 indicating the least amount of pain and 10 indicating the highest amount of pain. The pain interference items are each scored in the same way, but can also together generate an average score, with the minimum average score then being 0 and the maximum average score being 10. A higher score indicates a higher level of pain interference. Administered twice daily for 42 days.
Patient Health Questionnaire-2 (PHQ-2) | Six weeks
  A two-item version of the PHQ-9 made for assessing the level of interest and pleasure of doing things and, depression and hopelessness. The items are scored from 0 to 10. The minimum score is 0 and the maximum score is 20. Higher scores indicate higher levels of depression. Administered twice daily for 42 days.
Multidimensional Psychological Flexibility Inventory (MPFI) - Psychological Inflexibility | Six weeks
  Six items from the MPFI measuring psychological inflexibility. Assessing the domains; experiential avoidance, lack of contact with the present moment, self as content, fusion, lack of contact with values, and inaction. The items are scored from 0 to 10. The minimum score is 0 and the maximum score is 10. A higher average score indicates higher psychological inflexibility. Administered twice daily for 42 days.
Pain Catastrophizing Scale (PCS) | Six weeks
  Three items from the PCS measuring the level of catastrophizing when in pain. The items are scored from 0 to 10. The minimum score is 0 and the maximum score is 30. Higher scores indicate higher levels of pain catastrophizing. Administered twice daily for 42 days.
Weekly events | Six weeks
  A three-item measure developed by the research team to measure how the week has been in general, if something out of the ordinary has happened, and what this event was related to. The first item is from -10 to 10, with a higher score indicating a good week. The second item has five options and the third item has eight options for the participant to choose from. No summary score will be calculated, items are scored individually. Administered once a week for six weeks.
End of study questionnaire | Once approximately six weeks after intake
  An eight-item questionnaire developed by the research team assessing whether participants have begun any new treatment for their chronic pain condition, whether something out of the ordinary has happened during their study participation, and six items providing an opportunity for participants to give feedback on the study procedure, questionnaires, and platforms used in the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Department of Psychology, Uppsala University, Uppsala, Uppland, Sweden